CLINICAL TRIAL: NCT03267433
Title: A Randomized Phase III Trial of Consolidation With Autologous Hematopoietic Cell Transplantation Followed by Maintenance Rituximab vs Maintenance Rituximab Alone for Patients With Mantle Cell Lymphoma in Minimal Residual Disease-Negative First Complete Remission
Brief Title: Rituximab With or Without Stem Cell Transplant in Treating Patients With Minimal Residual Disease-Negative Mantle Cell Lymphoma in First Complete Remission
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA4151; NCI-2016-01403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA4151 (Other: ECOG-ACRIN Cancer Research Group); EA4151 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Stem Cell Transplantation; Specimen Handling; Fluid Therapy; Biopsy; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (auto-HCT, rituximab) (Experimental): Patients receive standard of care preparative chemotherapy and undergo auto-HCT. Beginning 100-140 days after transplant, patients receive rituximab IV or rituximab and hyaluronidase human SC or any approved rituximab biosimilar at the approved dose once every 8 weeks for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET, CT or PET/CT throughout the study. Patients may undergo blood sample collection during screening and on study. Patients also may undergo bone marrow biopsy and aspirate during screening.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human
- Group II (rituximab) (Experimental): Patients receive standard of care induction chemotherapy. Beginning 40-180 days after completion of chemotherapy, patients receive rituximab or rituximab and hyaluronidase human or any approved rituximab biosimilar at the approved dose, as in Group I. Patients undergo PET, CT or PET/CT throughout the study. Patients may undergo blood sample collection during screening and on study. Patients also may undergo bone marrow biopsy and aspirate during screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo HCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
  Arms: Group I (auto-HCT, rituximab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow biopsy and aspirate
  Other Names: BONE MARROW, LIQUID; Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspirate
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET or PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human

SUMMARY:
This phase III trial studies rituximab after stem cell transplant and to see how well it works compared with rituximab alone in treating patients with in minimal residual disease-negative mantle cell lymphoma in first complete remission. Immunotherapy with rituximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving chemotherapy before a stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving rituximab with or without stem cell transplant may work better in treating patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival in mantle cell lymphoma (MCL) patients in minimal residual disease (MRD)-negative first complete remission (CR) who undergo autologous hematopoietic stem cell transplantation (auto-HCT) followed by maintenance rituximab versus (vs.) maintenance rituximab alone (without auto-HCT).

SECONDARY OBJECTIVES:

I. To compare progression-free survival in MCL patients in MRD-negative CR who undergo auto-HCT followed by maintenance rituximab vs. maintenance rituximab alone.

II. To define the overall survival and progression-free survival at 2 and 5 years of chemosensitive but MRD-positive CR patients who undergo auto-HCT followed by 3 years of maintenance rituximab.

III. To define the overall survival and progression-free survival at 2 and 5 years of chemosensitive but MRD-positive partial response (PR) patients who undergo auto-HCT followed by 3 years of maintenance rituximab.

IV. To define the overall survival and progression-free survival at 2 and 5 years of MRD-negative PR patients who undergo auto-HCT followed by 3 years of maintenance rituximab.

V. To define the overall survival and progression-free survival at 2 and 5 years of MRD-indeterminate patients who undergo auto-HCT followed by 3 years of maintenance rituximab.

VI. To describe the rate of complications (serious infection, hospitalization, need for intravenous immune globulin) in MCL patients undergoing maintenance rituximab following auto-HCT.

VII. To determine the prognostic impact of MRD status at day 100, in MCL patients who were MRD-positive (including MRD-positive CR and MRD-positive PR) prior to auto-HCT.

EXPLORATORY TOBACCO USE OBJECTIVES:

I. To determine the effects of tobacco, operationalized as combustible tobacco (1a), other forms of tobacco (1b), and environmental tobacco exposure (ETS) (1c) on provider-reported cancer-treatment toxicity (adverse events (both clinical and hematologic) and dose modifications).

II. To determine the effects of tobacco on patient-reported physical symptoms and psychological symptoms.

III. To examine quitting behaviors and behavioral counseling/support and cessation medication utilization.

IV. To explore the effect of tobacco use and exposure on treatment duration, relative dose intensity, and therapeutic benefit.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive standard of care preparative chemotherapy and undergo auto-HCT. Beginning 100-140 days after transplant, patients receive rituximab intravenously (IV) or rituximab and hyaluronidase human subcutaneously (SC) or any approved rituximab biosimilar at the approved dose once every 8 weeks for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive standard of care induction chemotherapy. Beginning 40-180 days after completion of chemotherapy, patients receive rituximab or rituximab and hyaluronidase human or any approved rituximab biosimilar at the approved dose, as in Group I.

Patients undergo positron emission tomography (PET), computed tomography (CT) or PET/CT throughout the study. Patients may undergo blood sample collection during screening and on study. Patients also may undergo bone marrow biopsy and aspirate during screening.

After completion of study treatment, patients are followed up every 3 and 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR SCREENING (STEP 0 - PREREGISTRATION)
* Age >= 18 and =< 70 years
* Patients must have histologically confirmed mantle cell lymphoma, with cyclin D1 by immunohistochemical stains and/or t(11;14) by cytogenetics or fluorescence in situ hybridization (FISH). If patient has cyclin D1 negative mantle cell lymphoma with classical morphology and an expression profile (including SOX11+) that is otherwise indistinguishable from mantle cell lymphoma, communication with investigator is required for consideration of enrollment. The proliferation rate, using Ki-67 or MIB-1, should also be determined, but is not required until step 1 registration; patients may register to step 0 without a documented Ki-67 index
* In the opinion of the enrolling physician, patients must be felt to be a candidate for autologous stem cell transplantation
* Patient may be about to begin, be receiving or have completed induction therapy within 120 days prior to preregistration to step 0; no more than 300 days may have passed between the first day of induction therapy and preregistration to step 0

  * For patients who have completed induction therapy and have been restaged, restaging evaluation must show status of partial (PR) or complete response (CR); post-induction patients with evidence of clinical disease progression are not eligible for preregistration
  * Up to two regimens of therapy (conventional chemotherapy, antibody therapy, or an oral regimen) are allowed as long as a continuous response was ongoing throughout therapy; overall, a partial response needs to have been achieved (using studies at the time of diagnosis as the baseline)

    * NOTE: For example, a patient who started treatment with rituximab/bendamustine and was then switched to rituximab(R)-cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (CHOP) (due to insufficient response or excessive toxicity) would be counted as having received 2 regimens; however, R-CHOP alternating with R-dexamethasone, high-dose cytarabine, and cisplatin (DHAP) as a planned induction regimen would count as one regimen
* Patient does not have any documented history of central nervous system (CNS) involvement by mantle cell lymphoma; this includes no evidence of parenchymal brain, spinal cord, or cerebrospinal fluid involvement; radiculopathy symptoms from nerve root compression by lymphoma do not constitute CNS involvement
* Patient must have archived formalin-fixed paraffin-embedded (FFPE) tumor tissue specimen from the original diagnostic biopsy available for submission to Adaptive Biotechnologies for ClonoSEQ ID molecular marker identification of unique clonal immunoglobulin deoxyribonucleic acid (DNA) sequence

  * NOTE: If adequate tumor tissue is not available, peripheral blood collected prior to start of treatment with high disease burden (> 5%) is acceptable for molecular marker identification (ID) testing

    * Adaptive Biotechnologies will forward results within fourteen (14) days of receipt of any stored (e.g. frozen or FFPE) tumor tissue specimen to the submitting institution and to the ECOG-American College of Radiology Imaging Network (ACRIN) Operations Office
  * NOTE: Patients for whom the molecular marker is identified will have peripheral blood collected after completion of induction (patient's disease status is PR or CR) and submitted to Adaptive Biotechnologies for minimal residual disease (MRD) assessment

    * Adaptive Biotechnologies will forward results within ten to fourteen (10-14) days of receipt of fresh peripheral blood specimen to the submitting institution and to the ECOG-ACRIN Operations Office
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patients must have met eligibility criteria for the screening step 0
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): The proliferation rate, using Ki-67 or MIB-1 immunohistochemistry (=< 30% versus > 30% versus "indeterminate" Ki-67 index), must be documented for a baseline tumor biopsy specimen
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Institution has received results from Adaptive Biotechnologies as defined by one of the following criteria:

  * Patients are "MRD Indeterminate": ClonoSEQ ID molecular marker assessment did not identify any unique clonal immunoglobulin DNA sequence OR
  * ClonoSEQ ID molecular marker assessment identified unique clonal immunoglobulin DNA sequence and MRD assessment is completed
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patients must have completed induction therapy within 150 days prior to registration to step 1, AND no more than 300 days may have elapsed from the first dose of induction chemotherapy (cycle 1 [C1] day 1 [D1]) given, until the last day of induction chemotherapy administered; for those assigned to Arms A, C, or D, the date of transplant ("day 0") must not be greater than 365 days after the first dose of induction chemotherapy (C1D1) given

  * Patient must have received at least four (4) cycles of induction therapy
  * Up to two regimens of therapy (conventional chemotherapy, antibody therapy, or an oral regimen) are allowed as long as a continuous response was ongoing throughout therapy

    * NOTE: For example, a patient who started treatment with rituximab/bendamustine and was then switched to R-CHOP (due to insufficient response or excessive toxicity) would be counted as having received 2 regimens; however, R-CHOP alternating with R-DHAP as a planned induction regimen would count as one regimen
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patients must have achieved a radiologic complete or partial remission as defined by the Lugano criteria
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): In the opinion of the enrolling physician, patients must be felt to be a candidate for autologous stem cell transplantation
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patients have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Human immunodeficiency virus (HIV) positive patients are not excluded, but to enroll, must meet all of the below criteria:

  * HIV is sensitive to antiretroviral therapy
  * Must be willing to take effective antiretroviral therapy that has minimal overlapping toxicity and pharmacokinetic interactions with protocol therapy
  * No history of HIV-related opportunistic disease or acquired immune deficiency syndrome (AIDS)-defining conditions within past 12 months other than historic CD4+ T-cell counts below 200 cells/mm^3
  * Expected long-term survival if lymphoma were not present
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patient must be disease-free >= 3 years of prior malignancies with the exception of adequately treated non-melanoma skin cancer, adequately treated in situ carcinoma, melanoma in situ post wide local excision or Mohs surgery, low grade prostate carcinoma (Gleason grade =< 6) managed with observation that has been stable for at least 6 months
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patient must not be pregnant or breast-feeding due to the potential for congenital abnormalities and of harm to nursing infants due to the treatment regimens used

  * All patients of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
  * A patient of childbearing potential is anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* INCLUSION CRITERIA FOR TREATMENT ASSIGNMENT (STEP 1): Patient of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study and for 12 months post rituximab treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in mantle cell lymphoma (MCL) patients in minimal residual disease (MRD)-negative complete remission (CR) who undergo auto-hematopoietic stem cell transplant (HCT) followed by rituximab versus (vs.) maintenance rituximab alone | Time between randomization and death from any cause, assessed up to 10 years
  The Kaplan-Meier method will be used to estimate OS, including medians and confidence intervals. Comparison of OS between treatment arms will be conducted using a one-sided log-rank test stratified with mantle cell lymphoma International Prognostic Index (MIPI)-c score and induction regimen.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in MCL patients in MRD-negative CR who undergo auto-HCT followed by rituximab vs rituximab alone | From randomization to the earliest of documented disease progression or death without progression, assessed up to 10 years
  The method of Kaplan and Meier will be used to estimate PFS, and stratified log-rank test will be used to compare PFS between two arms.
PFS in MRD-negative PR patients, MRD-positive CR patients, MRD-positive PR patients, and MRD-indeterminate patients who undergo auto-HCT followed by rituximab | From randomization to the earliest of documented disease progression or death without progression, assessed up to 10 years
  Will be estimated by the method of Kaplan and Meier.
OS in MRD-negative PR patients, MRD-positive CR patients, MRD-positive PR patients, and MRD-indeterminate patients who undergo auto-HCT followed by rituximab | Time between randomization and death from any cause, assessed up to 10 years
  Will be estimated by the method of Kaplan and Meier.
Rate of complications in MCL patients undergoing maintenance rituximab | Up to 10 years
MRD status in MCL patients who were MRD-positive prior to auto-HCT | At 100 days after HCT
  Conversion rate will be reported together with confidence intervals.
Incidence of adverse events | Up to 10 years
  Will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The primary safety analysis will be based on the toxicity population, and the analysis will be performed by treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Fenske, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (375):
- United States (374):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Stateville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Kumar A. What is the role of up-front autologous stem cell transplantation in mantle cell lymphoma? Hematology Am Soc Hematol Educ Program. 2022 Dec 9;2022(1):155-162. doi: 10.1182/hematology.2022000333. PMID 36485104
- [Derived] Thiruvengadam SK, Hunter B, Varnavski A, Fakhri B, Kaplan L, Ai WZ, Pampaloni M, Huang CY, Martin T 3rd, Damon L, Andreadis CB. Ofatumumab, Etoposide, and Cytarabine Intensive Mobilization Regimen in Patients with High-risk Relapsed/Refractory Diffuse Large B-Cell Lymphoma Undergoing Autologous Stem Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):246-256.e2. doi: 10.1016/j.clml.2020.11.005. Epub 2020 Nov 11. PMID 33288485